CLINICAL TRIAL: NCT06639282
Title: SIPO1-AD: A Phase II Clinical Trial for the Assessment of Safety, Tolerability, and Efficacy of Siponimod in Patients With Mild Alzheimer&Amp;#39;s Disease Dementia
Brief Title: Repurposing Siponimod for Alzheimer's Disease
Acronym: SIPO1-AD
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Collaborators: Texas Tech University Health Sciences Center (Other); Arizona State University (Other); National Institute on Aging (NIA) (NIH); Novartis (Industry); Laboratory Corporation of America (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 23-500-037-10-03; 7R01AG073212-02 (NIH)
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Alzheimer Disease; Mild Alzheimer Disease; MCI With Increased Risk for Alzheimer Disease; Cognitive Impairment, Mild
Keywords: Alzheimer's disease; Siponimod; Cognitive Impairment; Cognition; Brain Imaging; Biomarkers; Immunomodulation
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — siponimod

STUDY DESIGN:
Intervention Model Description: The study will have 105 participants with a 2:1 ratio of drug:placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The clinical research coordinator, the psychometrist, the co-investigators (Dr. Boris Decourt and Dr. Karl Golnik) will be masked. Everyone who is patient-facing will be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Drug Arm (Experimental): Randomly assigned subjects who will receive an escalating dose of Siponimod (0.25-1 mg/day) for 12 months.
  Interventions: Drug: Siponimod
- Placebo Arm (Placebo Comparator): Randomly assigned subjects who will receive a placebo daily for 12 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Siponimod — Siponimod (formerly known as BAF312 and completed trial NCT #01665144) has been FDA approved since 2019 (IND #076122) for the treatment of multiple sclerosis. Siponimod is an immunomodulator that prevents the egression of T lymphocytes from peripheral lymphoid organs.
  Other Names: Mayzent
  Arms: Drug Arm
Drug: Placebo — A placebo that resembles siponimod will be given once daily to participants randomly assigned into the placebo arm.
  Arms: Placebo Arm

SUMMARY:
Collaboration with multiple sclerosis (MS) specialty colleagues led us to formulate the central hypothesis that Siponimod could lower the rate of brain atrophy in Alzheimer's disease (AD) subjects. To test our central hypothesis, we will carry out an 18-month Phase II, double-blind, randomized, twoarmed, placebo controlled, proof-of-concept clinical study in early AD subjects (i.e. mild AD) who will be receiving an escalating dose of Siponimod or placebo in the ratio 2:1 for 12 months, followed by a 6-month washout period. The primary outcome measures are safety and tolerability of Siponimod in mild AD subjects. The secondary outcome measures are the rates of brain atrophy derived from volumetric MRI (vMRI) as a proxy for neurodegeneration conducted at baseline, 6, 12, and 18 months. The tertiary outcome measures are the changes in cognition and the levels of AD-associated (e.g., Aβ and tau) and inflammatory biomarkers in CSF after Siponimod exposure. In an exploratory effort, we will also measure plasma inflammatory markers during the entire duration of the study to investigate whether one or more of these markers can be used as dynamic surrogate markers of treatment response. Using our unique experience with the repurposing of immunomodulatory drugs for AD (and NCT #04032626), in the present project we are using elements of clinical trial design that we believe were successful and made some adjustments to fit the pharmacologic and toxic properties of Siponimod.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is a neurodegenerative disorder with several complex neuropathologies suspected to develop sequentially but that overlap over time as symptoms progress to dementia. Thus, to be effective, future intervention strategies will likely require combination therapies or pleiotropic agents to tackle several AD molecular pathogenic pathways simultaneously. For more than a decade, our group has been exploring the repurposing of immunomodulators for AD. Recent discussions with collaborators who specialize in multiple sclerosis suggest that sphingosine-1-phosphate receptor (S1PR) modulators are strong candidates for repurposing in AD. Indeed, S1PR modulators are blood brain barrier (BBB) penetrant and display pleiotropic actions, including immunomodulation and neuroprotective properties. S1P is a versatile endogenous molecule that regulates several signaling pathways by binding to five G-protein-coupled receptors, which are expressed in high levels in cardiac, vascular, immune, and brain cells. This widespread localization of S1PR was the historical basis for Novartis Pharmaceuticals, Inc, to develop oral formulations of S1PR modulators for multiple sclerosis (MS), which proved successful and resulted in two marketed oral compounds (i.e., fingolimod and Siponimod). In the present project, we intend to collaborate with Novartis to use the most recently FDA-approved S1PR modulator, Siponimod. Based on MS and animal experimentation literature, we hypothesize that Siponimod could alter the rate of neurodegeneration as measured by lowering the rate of brain atrophy in mild AD dementia subjects. In this Phase II, proof-of-concept, translational clinical study, mild AD dementia subjects will be randomized 2:1 and will receive gradual titration regimen of Siponimod starting at 0.25mg/day and increasing up to final dosage of 1 mg/day (N=70) or placebo (N=35) for 12 months. This will be followed by a 6-month washout period. Siponimod has demonstrated positive immunomodulatory and neuroprotective actions in MS patients, and because its toxicity profile is favorable for use in older individuals, Siponimod has a strong potential to alter markers of mild AD dementia pathology and disease trajectory.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female at least 50 years of age, but less than 85 (84 at time of screening)
2. Females must be of non-childbearing potential or have negative pregnancy test at time of screening. Women of non-childbearing potential are defined as women who are either permanently sterilized (hysterectomy, bilateral oophorectomy or bilateral salpingectomy) or who are postmenopausal. Women will be considered postmenopausal if they have been amenorrheic for >=12 months prior to the planned date of enrollment.
3. Must have a diagnosis of mild Alzheimer's Dementia determined by medical record review.
4. Vision and hearing must be sufficient to comply with study procedures. Be able to take oral medications.
5. Must be able to attend all study visits indicated in the schedule of visits.
6. Must have a collateral informant/study partner who has significant direct contact with the patient at least 10 hours per week and who is willing to accompany the patient to specified clinic visits, supervise administration of all study medication, and be available for telephone visits/interviews.
7. Documented Mini Mental State Exam (MMSE) score between 21-26 at Screening Visit.
8. CT or MRI scan of the brain within 12 months of enrollment showing no evidence of significant focal lesions or other pathology which could contribute to dementia. If neither a CT nor an MRI scan is available from the past 12 months, a CT scan fulfilling the requirements must be obtained before randomization.
9. Hachinski ischemic score must be < 4.
10. Geriatric depression scale must be < 10.
11. Prior to dosing all randomized study subjects must show proof they have received immunization to varicella (VZV IgG).
12. If the patient has a legally authorized representative (LAR), the LAR must review and sign the informed consent form. If the patient does not have a LAR, the patient must appear able to provide informed consent and must review and sign the informed consent form. In addition, the patient's informant/study partner (as defined above) must sign an informed consent form. If the LAR and the patient's informant /study partner are the same individual, he/she should sign under both designations.

Exclusion Criteria:

1. Taking one of the following medications: Medications for treatment of cancer or other drugs that weaken the immune system (ex. Natalizumab and Rituximab), Amiodarone, Bishydroxycoumarin, Chloramphenicol, Cimetidine, Fluconazole, Fluvastatin, Miconazole, Phenylbutazone, Sulphinpyrazone, Sulphadiazine, Sulphamethizole, Sulfamethoxazole, Sulphaphenazole, Trimethoprim, and Zafirlukast.
2. Current active infection in participants including, but not limited to, herpes zoster, herpes infection, bronchitis, sinusitis, upper respiratory infection and fungal skin infection. Siponimod may increase the risk in participants with active infections.
3. If participant received mRNA COVID-19 vaccination, must have received last dose at least 3 months prior to first dose of study drug/placebo.
4. Current evidence or history within the last 3 years of a neurological or psychiatric illness that could contribute to dementia, including (but not limited to) epilepsy, focal brain lesion, Parkinson's disease, seizure disorder, or head injury with loss of consciousness.
5. Meets DSM IV criteria for any major psychiatric disorder including psychosis, major depression and bipolar disorder.
6. Known history of self-reported alcohol and/ or substance abuse.
7. Isolated living circumstances which would prohibit a study partner from providing sufficient and credible information about the participant.
8. Poorly controlled hypertension
9. Known Atrioventricular heart block, known heart block type I-III.
10. History of myocardial infarction or signs or symptoms of unstable coronary artery disease within the last year (including revascularization procedure/angioplasty).
11. Severe pulmonary disease (including chronic obstructive pulmonary disease) requiring more than 2 hospitalizations within the past year.
12. Untreated obstructive sleep apnea.
13. Any thyroid disease (unless euthyroid on treatment for at least 6 months prior to screening). [15] Active neoplastic disease (except for skin tumors other than melanoma). Patients with a history of prior malignancy are eligible provided they were treated with curative intent and (i) do not require any longer any active therapy; (ii) being considered in complete remission; and (iii) after the Medical Monitor's assessment/approval of each case.
14. Prior prostate cancer or new diagnosis of prostate cancer.
15. History of multiple myeloma.
16. Absolute lymphocytopenia of <1,000/mm3, or a history of lymphocytopenia.
17. Absolute neutropenia of <1,000/mm3, or a history of neutropenia.
18. History of/ or current thromboembolism (including deep venous thrombosis).
19. Any clinically significant hepatic or renal disease (including presence of Hepatitis B or C surface antigen or an elevated transaminase levels of greater than 2x the upper limit of normal (ULN) or creatinine greater than 1.5 x upper limit of normal (ULN)).
20. Clinically significant hematologic or coagulation disorder including any unexplained anemia, or a platelet count less than 100,000/μL at screening.
21. Use of any investigational drug within 30 days or within five half-lives of the investigational agent, whichever is longer.
22. Unwilling or unable to undergo CT or MRI imaging.
23. In the opinion of the investigator, participation would not be in the best interest of the subject.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2029-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Monitoring and recording of all adverse events (AEs) and serious adverse events (SAEs) | 18 months
  To evaluate the safety and tolerability of Siponimod titrated for up to 12 months and washed out for 6 months in mild AD subjects. (Subjects will receive gradual titration regimen of Siponimod starting at 0.25mg/day and increasing every two weeks by 0.25 mg, up to final dosage of 1 mg/day.) Safety will be assessed at each study visit through completion of comprehensive tests and procedures aimed at monitoring for potentials adverse events (AEs). Study staff will also gather direct reports from subjects regarding any adverse events.

SECONDARY OUTCOMES:
Rates of brain atrophy | 12 months
  The secondary outcome measures are the rates of brain atrophy derived from volumetric MRI (vMRI) as a proxy for neurodegeneration conducted at baseline. The aim is to assess the medical benefits of the drug in mild AD dementia subjects by assessing whether brain atrophy slows with Siponimod treatment 1 mg/day titrated for up to 12 months. (Subjects will receive gradual titration regimen of Siponimod starting at 0.25mg/day and increasing every two weeks by 0.25 mg, up to final dosage of 1 mg/day.)
  Subjects will undergo volumetric MRI (vMRI) measurements of the hippocampus, cortical thickness, and global thickness as indicators of neurodegeneration.

OTHER OUTCOMES:
Changes in cognition assessed by Mini Mental State Examination (MMSE) | 18 months
  To evaluate how siponimod 1 mg/day titrated for up to 12 months and washed out for 6 months affects changes in cognition assessed by the Mini Mental State Examination (MMSE). (Subjects will receive gradual titration regimen of Siponimod starting at 0.25mg/day and increasing every two weeks by 0.25 mg, up to final dosage of 1 mg/day.) MMSE Scores range from 0 to 30, with 30 being the score assigned to cognitively normal individuals. The range for mild AD is 21-26. A higher score is better.
Changes in cognition as assessed by Alzheimer's Disease Composite Score (ADCOMS) | 18 months
  To evaluate the effect on cognition Alzheimer's Disease Composite Score (ADCOMS) of siponimod 1mg/day titrated for up to 12 months and washed out for 6 months. (Subjects will receive gradual titration regimen of Siponimod starting at 0.25mg/day and increasing every two weeks by 0.25 mg, up to final dosage of 1 mg/day.) The lowest ADCOMS score is 0, while the highest is 1.97. A lower score is better.
Changes in cognition assessed by Alzheimer's Disease Assessment Scale - Cognitive (ADAS-cog) | 18 months
  To evaluate how siponimod 1 mg/day titrated for up to 12 months and washed out for 6 months affects changes in cognition assessed by the Alzheimer's Disease Assessment Scale - Cognitive (ADAS-cog) assessment. (Subjects will receive gradual titration regimen of Siponimod starting at 0.25mg/day and increasing every two weeks by 0.25 mg, up to final dosage of 1 mg/day.) A higher ADAS-cog score indicates more impairment; the range is 0 to 89.
Changes in cognition assessed by Clinical Dementia Rating - Sum of Boxes (CDR-SOB) | 18 months
  To evaluate how siponimod 1 mg/day titrated for up to 12 months and washed out for 6 months affects changes in cognition assessed by the Clinical Dementia Rating - Sum of Boxes (CDR-SOB) test. (Subjects will receive gradual titration regimen of Siponimod starting at 0.25mg/day and increasing every two weeks by 0.25 mg, up to final dosage of 1 mg/day.)
  The CDR-SOB ratings of degree of impairment obtained on each of the 6 categories of function are synthesized into one global rating of dementia (ranging from 0 to 3). A score of 0 indicates no dementia, while higher scores indicate increasingly higher levels of dementia.
Changes in cognition assessed by Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS-ADL) | 18 months
  To evaluate how siponimod 1 mg/day titrated for up to 12 months and washed out for 6 months affects changes in cognition assessed by the Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS-ADL) assessment. (Subjects will receive gradual titration regimen of Siponimod starting at 0.25mg/day and increasing every two weeks by 0.25 mg, up to final dosage of 1 mg/day.) The ADCS-ADL assessment score range is 0-78. A higher score is better.
Plasma inflammatory markers | 18 months
  In an exploratory effort, we will also measure plasma inflammatory markers to evaluate the effect on blood inflammatory markers (plasma C-reactive protein, TNF-a, IL-1B, IL-6, IL-8, and IL-10) of siponimod 1 mg/day titrated for up to 12 months and washed out for 6 months. (Subjects will receive gradual titration regimen of Siponimod starting at 0.25mg/day and increasing every two weeks by 0.25 mg, up to final dosage of 1 mg/day.)
Saliva biomarkers | 18 months
  To evaluate the effect of siponimod 1 mg/day titrated for up to 12 months and washed out for 6 months on Saliva markers AB40 and AB2. (Subjects will receive gradual titration regimen of Siponimod starting at 0.25mg/day and increasing every two weeks by 0.25 mg, up to final dosage of 1 mg/day.)
Cerebrospinal fluid biomarkers | 12 months
  To evaluate the effect of siponimod 1 mg/day titrated for up to 12 months on the levels of AD-associated (e.g., Aβ and tau) and inflammatory biomarkers in cerebrospinal fluid (CSF). CSF biomarkers that will be assessed include amyloid beta 40 and 42, Tau, and Phospo-Tau, CSF C-reactive protein, TNF-a, IL-1B, IL-6, IL8, and IL-10. (Subjects will receive gradual titration regimen of Siponimod starting at 0.25mg/day and increasing every two weeks by 0.25 mg, up to final dosage of 1 mg/day.)

CONTACTS AND LOCATIONS:
Overall Officials: Marwan N Sabbagh, MD, Principal Investigator — St. Joseph's Hospital and Medical Center, Phoenix; Boris Decourt, PhD, Study Chair — Texas Tech University Health Sciences Center
Locations (1):
- St. Joseph's Hospital and Medical Center, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
Information from the study such as SAEs, the study protocol, case report forms, study results, Statistical Analysis Plan, Informed Consent Form, and findings that might alter the current benefit-risk profile of the Study Drug or that would be sufficient to consider changes in the Study Drug's administration or in the overall conduct of the Study, and the Clinical Study Report, will be shared with the drug manufacturer Novartis, and the subaward institutions, Arizona State University and Texas Tech, and the members of the Data Safety and Monitoring Board, who are associated with University of Indiana, Pentara Corporation, and Texas Tech, and the internal medical monitor and clinical monitoring team who are part of Barrow Neurological Institute (BNI).
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: From 03/08/2023 to 07/31/2027
Access Criteria: Dr. Jeffrey Wilson at Arizona State University will be given study data directly from Barrow Neurological Institute (BNI) staff to perform biostatistical analysis. Dr. Boris Decourt at Texas Tech will be given blood and saliva samples from BNI to process, store, and analyze. Dr. Mirla Avila at Texas Tech, Dr. Martin Farlow at University of Indiana, and Dr. Craig Mallinckrodt at Pentara Corporation will receive case report forms from BNI staff such as the project manager and SAE information from Dr. Sabbagh. There are current data use and material transfer agreements in place with the respective institutions. Dr. Sabbagh and Dr. Decourt also plan to present study findings in the form of peer-reviewed manuscripts and presentations at scientific meetings.

REFERENCES:
- [Background] Kahle-Wrobleski K, Coley N, Lepage B, Cantet C, Vellas B, Andrieu S; Plasa DSA Group. Understanding the complexities of functional ability in Alzheimer's disease: more than just basic and instrumental factors. Curr Alzheimer Res. 2014 May;11(4):357-66. doi: 10.2174/1567205011666140317101419. PMID 24635843
- [Background] Morris JC, Storandt M, Miller JP, McKeel DW, Price JL, Rubin EH, Berg L. Mild cognitive impairment represents early-stage Alzheimer disease. Arch Neurol. 2001 Mar;58(3):397-405. doi: 10.1001/archneur.58.3.397. PMID 11255443
- [Background] Tahami Monfared AA, Houghton K, Zhang Q, Mauskopf J; Alzheimer's Disease Neuroimaging Initiative. Staging Disease Severity Using the Alzheimer's Disease Composite Score (ADCOMS): A Retrospective Data Analysis. Neurol Ther. 2022 Mar;11(1):413-434. doi: 10.1007/s40120-022-00326-y. Epub 2022 Jan 31. PMID 35099758
- [Background] Decourt B, Wilson J, Ritter A, Dardis C, DiFilippo FP, Zhuang X, Cordes D, Lee G, Fulkerson ND, St Rose T, Hartley K, Sabbagh MN. MCLENA-1: A Phase II Clinical Trial for the Assessment of Safety, Tolerability, and Efficacy of Lenalidomide in Patients with Mild Cognitive Impairment Due to Alzheimer's Disease. Open Access J Clin Trials. 2020;12:1-13. doi: 10.2147/oajct.s221914. Epub 2020 Jan 7. PMID 32123490
- [Background] Wang J, Logovinsky V, Hendrix SB, Stanworth SH, Perdomo C, Xu L, Dhadda S, Do I, Rabe M, Luthman J, Cummings J, Satlin A. ADCOMS: a composite clinical outcome for prodromal Alzheimer's disease trials. J Neurol Neurosurg Psychiatry. 2016 Sep;87(9):993-9. doi: 10.1136/jnnp-2015-312383. Epub 2016 Mar 23. PMID 27010616
- [Background] Vassar R. BACE1 inhibitor drugs in clinical trials for Alzheimer's disease. Alzheimers Res Ther. 2014 Dec 24;6(9):89. doi: 10.1186/s13195-014-0089-7. eCollection 2014. PMID 25621019
- [Background] Tur C, Kalincik T, Oh J, Sormani MP, Tintore M, Butzkueven H, Montalban X. Head-to-head drug comparisons in multiple sclerosis: Urgent action needed. Neurology. 2019 Oct 29;93(18):793-809. doi: 10.1212/WNL.0000000000008319. Epub 2019 Oct 7. PMID 31591277
- [Background] Golde TE, Koo EH, Felsenstein KM, Osborne BA, Miele L. gamma-Secretase inhibitors and modulators. Biochim Biophys Acta. 2013 Dec;1828(12):2898-907. doi: 10.1016/j.bbamem.2013.06.005. Epub 2013 Jun 17. PMID 23791707
- [Background] Frost GR, Jonas LA, Li YM. Friend, Foe or Both? Immune Activity in Alzheimer's Disease. Front Aging Neurosci. 2019 Dec 10;11:337. doi: 10.3389/fnagi.2019.00337. eCollection 2019. PMID 31920620
- [Background] Yiannopoulou KG, Anastasiou AI, Zachariou V, Pelidou SH. Reasons for Failed Trials of Disease-Modifying Treatments for Alzheimer Disease and Their Contribution in Recent Research. Biomedicines. 2019 Dec 9;7(4):97. doi: 10.3390/biomedicines7040097. PMID 31835422
- [Background] Xie HG, Prasad HC, Kim RB, Stein CM. CYP2C9 allelic variants: ethnic distribution and functional significance. Adv Drug Deliv Rev. 2002 Nov 18;54(10):1257-70. doi: 10.1016/s0169-409x(02)00076-5. PMID 12406644
- [Background] Wyss-Coray T, Rogers J. Inflammation in Alzheimer disease-a brief review of the basic science and clinical literature. Cold Spring Harb Perspect Med. 2012 Jan;2(1):a006346. doi: 10.1101/cshperspect.a006346. PMID 22315714
- [Background] Shakeri-Nejad K, Aslanis V, Veldandi UK, Mooney L, Pezous N, Brendani B, Juan A, Allison M, Perry R, Legangneux E. Effects of Therapeutic and Supratherapeutic Doses of Siponimod (BAF312) on Cardiac Repolarization in Healthy Subjects. Clin Ther. 2015 Nov 1;37(11):2489-2505.e2. doi: 10.1016/j.clinthera.2015.09.006. Epub 2015 Oct 27. PMID 26519230
- [Background] Sabbagh MN, Shi J, Lee M, Arnold L, Al-Hasan Y, Heim J, McGeer P. Salivary beta amyloid protein levels are detectable and differentiate patients with Alzheimer's disease dementia from normal controls: preliminary findings. BMC Neurol. 2018 Sep 26;18(1):155. doi: 10.1186/s12883-018-1160-y. PMID 30257642
- [Background] Rosen WG, Mohs RC, Davis KL. A new rating scale for Alzheimer's disease. Am J Psychiatry. 1984 Nov;141(11):1356-64. doi: 10.1176/ajp.141.11.1356. PMID 6496779
- [Background] Peskind ER, Riekse R, Quinn JF, Kaye J, Clark CM, Farlow MR, Decarli C, Chabal C, Vavrek D, Raskind MA, Galasko D. Safety and acceptability of the research lumbar puncture. Alzheimer Dis Assoc Disord. 2005 Oct-Dec;19(4):220-5. doi: 10.1097/01.wad.0000194014.43575.fd. PMID 16327349
- [Background] Morris JC. The Clinical Dementia Rating (CDR): current version and scoring rules. Neurology. 1993 Nov;43(11):2412-4. doi: 10.1212/wnl.43.11.2412-a. No abstract available. PMID 8232972
- [Background] Mizutani T. PM frequencies of major CYPs in Asians and Caucasians. Drug Metab Rev. 2003 May-Aug;35(2-3):99-106. doi: 10.1081/dmr-120023681. PMID 12959412
- [Background] McKhann GM, Knopman DS, Chertkow H, Hyman BT, Jack CR Jr, Kawas CH, Klunk WE, Koroshetz WJ, Manly JJ, Mayeux R, Mohs RC, Morris JC, Rossor MN, Scheltens P, Carrillo MC, Thies B, Weintraub S, Phelps CH. The diagnosis of dementia due to Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):263-9. doi: 10.1016/j.jalz.2011.03.005. Epub 2011 Apr 21. PMID 21514250
- [Background] Mauri M, Sinforiani E, Zucchella C, Cuzzoni MG, Bono G. Progression to dementia in a population with amnestic mild cognitive impairment: clinical variables associated with conversion. Funct Neurol. 2012 Jan-Mar;27(1):49-54. PMID 22687167
- [Background] Martinez B, Peplow PV. Amelioration of Alzheimer's disease pathology and cognitive deficits by immunomodulatory agents in animal models of Alzheimer's disease. Neural Regen Res. 2019 Jul;14(7):1158-1176. doi: 10.4103/1673-5374.251192. PMID 30804241
- [Background] Limmroth V, Ziemssen T, Lang M, Richter S, Wagner B, Haas J, Schmidt S, Gerbershagen K, Lassek C, Klotz L, Hoffmann O, Albert C, Schuh K, Baier-Ebert M, Wendt G, Schieb H, Hoyer S, Dechend R, Haverkamp W. Electrocardiographic assessments and cardiac events after fingolimod first dose - a comprehensive monitoring study. BMC Neurol. 2017 Jan 18;17(1):11. doi: 10.1186/s12883-016-0789-7. PMID 28100182
- [Background] Leverenz JB, Raskind MA. Early amyloid deposition in the medial temporal lobe of young Down syndrome patients: a regional quantitative analysis. Exp Neurol. 1998 Apr;150(2):296-304. doi: 10.1006/exnr.1997.6777. PMID 9527899
- [Background] Legangneux E, Gardin A, Johns D. Dose titration of BAF312 attenuates the initial heart rate reducing effect in healthy subjects. Br J Clin Pharmacol. 2013 Mar;75(3):831-41. doi: 10.1111/j.1365-2125.2012.04400.x. PMID 22845008
- [Background] Lannfelt L, Moller C, Basun H, Osswald G, Sehlin D, Satlin A, Logovinsky V, Gellerfors P. Perspectives on future Alzheimer therapies: amyloid-beta protofibrils - a new target for immunotherapy with BAN2401 in Alzheimer's disease. Alzheimers Res Ther. 2014 Mar 24;6(2):16. doi: 10.1186/alzrt246. eCollection 2014. PMID 25031633
- [Background] Kappos L, Bar-Or A, Cree BAC, Fox RJ, Giovannoni G, Gold R, Vermersch P, Arnold DL, Arnould S, Scherz T, Wolf C, Wallstrom E, Dahlke F; EXPAND Clinical Investigators. Siponimod versus placebo in secondary progressive multiple sclerosis (EXPAND): a double-blind, randomised, phase 3 study. Lancet. 2018 Mar 31;391(10127):1263-1273. doi: 10.1016/S0140-6736(18)30475-6. Epub 2018 Mar 23. PMID 29576505
- [Background] Juif PE, Kraehenbuehl S, Dingemanse J. Clinical pharmacology, efficacy, and safety aspects of sphingosine-1-phosphate receptor modulators. Expert Opin Drug Metab Toxicol. 2016 Aug;12(8):879-95. doi: 10.1080/17425255.2016.1196188. Epub 2016 Jun 13. PMID 27249325
- [Background] Jack CR Jr, Knopman DS, Jagust WJ, Petersen RC, Weiner MW, Aisen PS, Shaw LM, Vemuri P, Wiste HJ, Weigand SD, Lesnick TG, Pankratz VS, Donohue MC, Trojanowski JQ. Tracking pathophysiological processes in Alzheimer's disease: an updated hypothetical model of dynamic biomarkers. Lancet Neurol. 2013 Feb;12(2):207-16. doi: 10.1016/S1474-4422(12)70291-0. PMID 23332364
- [Background] Jack CR Jr, Slomkowski M, Gracon S, Hoover TM, Felmlee JP, Stewart K, Xu Y, Shiung M, O'Brien PC, Cha R, Knopman D, Petersen RC. MRI as a biomarker of disease progression in a therapeutic trial of milameline for AD. Neurology. 2003 Jan 28;60(2):253-60. doi: 10.1212/01.wnl.0000042480.86872.03. PMID 12552040
- [Background] Heneka MT, Carson MJ, El Khoury J, Landreth GE, Brosseron F, Feinstein DL, Jacobs AH, Wyss-Coray T, Vitorica J, Ransohoff RM, Herrup K, Frautschy SA, Finsen B, Brown GC, Verkhratsky A, Yamanaka K, Koistinaho J, Latz E, Halle A, Petzold GC, Town T, Morgan D, Shinohara ML, Perry VH, Holmes C, Bazan NG, Brooks DJ, Hunot S, Joseph B, Deigendesch N, Garaschuk O, Boddeke E, Dinarello CA, Breitner JC, Cole GM, Golenbock DT, Kummer MP. Neuroinflammation in Alzheimer's disease. Lancet Neurol. 2015 Apr;14(4):388-405. doi: 10.1016/S1474-4422(15)70016-5. PMID 25792098
- [Background] Goodman AD, Anadani N, Gerwitz L. Siponimod in the treatment of multiple sclerosis. Expert Opin Investig Drugs. 2019 Dec;28(12):1051-1057. doi: 10.1080/13543784.2019.1676725. Epub 2019 Nov 3. PMID 31603362
- [Background] Gate D, Saligrama N, Leventhal O, Yang AC, Unger MS, Middeldorp J, Chen K, Lehallier B, Channappa D, De Los Santos MB, McBride A, Pluvinage J, Elahi F, Tam GK, Kim Y, Greicius M, Wagner AD, Aigner L, Galasko DR, Davis MM, Wyss-Coray T. Clonally expanded CD8 T cells patrol the cerebrospinal fluid in Alzheimer's disease. Nature. 2020 Jan;577(7790):399-404. doi: 10.1038/s41586-019-1895-7. Epub 2020 Jan 8. PMID 31915375
- [Background] Gaser C, Franke K, Kloppel S, Koutsouleris N, Sauer H; Alzheimer's Disease Neuroimaging Initiative. BrainAGE in Mild Cognitive Impaired Patients: Predicting the Conversion to Alzheimer's Disease. PLoS One. 2013 Jun 27;8(6):e67346. doi: 10.1371/journal.pone.0067346. Print 2013. PMID 23826273
- [Background] Gardin A, Ufer M, Legangneux E, Rossato G, Jin Y, Su Z, Pal P, Li W, Shakeri-Nejad K. Effect of Fluconazole Coadministration and CYP2C9 Genetic Polymorphism on Siponimod Pharmacokinetics in Healthy Subjects. Clin Pharmacokinet. 2019 Mar;58(3):349-361. doi: 10.1007/s40262-018-0700-3. PMID 30088221
- [Background] Galasko D, Bennett D, Sano M, Ernesto C, Thomas R, Grundman M, Ferris S. An inventory to assess activities of daily living for clinical trials in Alzheimer's disease. The Alzheimer's Disease Cooperative Study. Alzheimer Dis Assoc Disord. 1997;11 Suppl 2:S33-9. PMID 9236950
- [Background] Fox R, Arnold D, Giovannoni G, Cree B, Vermersch P, Bar-Or A, Gold R, Benedict R, Meier DP, Arnould S, Ritter S, Dahlke F, Karlsson G, Kappos L (2020) Siponimod Reduces Grey Matter Atrophy in Patients with Secondary Progressive Multiple Sclerosis: Subgroup Analyses from the EXPAND Study (1130). Neurology 94:1130.
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Elmaleh DR, Farlow MR, Conti PS, Tompkins RG, Kundakovic L, Tanzi RE. Developing Effective Alzheimer's Disease Therapies: Clinical Experience and Future Directions. J Alzheimers Dis. 2019;71(3):715-732. doi: 10.3233/JAD-190507. PMID 31476157
- [Background] Derfuss T, Mehling M, Papadopoulou A, Bar-Or A, Cohen JA, Kappos L. Advances in oral immunomodulating therapies in relapsing multiple sclerosis. Lancet Neurol. 2020 Apr;19(4):336-347. doi: 10.1016/S1474-4422(19)30391-6. Epub 2020 Feb 11. PMID 32059809
- [Background] Decourt B, Drumm-Gurnee D, Wilson J, Jacobson S, Belden C, Sirrel S, Ahmadi M, Shill H, Powell J, Walker A, Gonzales A, Macias M, Sabbagh MN. Poor Safety and Tolerability Hamper Reaching a Potentially Therapeutic Dose in the Use of Thalidomide for Alzheimer's Disease: Results from a Double-Blind, Placebo-Controlled Trial. Curr Alzheimer Res. 2017;14(4):403-411. doi: 10.2174/1567205014666170117141330. PMID 28124585
- [Background] De Stefano N, Silva DG, Barnett MH. Effect of Fingolimod on Brain Volume Loss in Patients with Multiple Sclerosis. CNS Drugs. 2017 Apr;31(4):289-305. doi: 10.1007/s40263-017-0415-2. PMID 28247239
- [Background] Crivelli SM, Giovagnoni C, Visseren L, Scheithauer AL, de Wit N, den Hoedt S, Losen M, Mulder MT, Walter J, de Vries HE, Bieberich E, Martinez-Martinez P. Sphingolipids in Alzheimer's disease, how can we target them? Adv Drug Deliv Rev. 2020;159:214-231. doi: 10.1016/j.addr.2019.12.003. Epub 2020 Jan 3. PMID 31911096
- [Background] Bordet R, Camu W, De Seze J, Laplaud DA, Ouallet JC, Thouvenot E. Mechanism of action of s1p receptor modulators in multiple sclerosis: The double requirement. Rev Neurol (Paris). 2020 Jan-Feb;176(1-2):100-112. doi: 10.1016/j.neurol.2019.02.007. Epub 2019 Nov 19. PMID 31757428
- [Background] Bigaud M, Rudolph B, Briard E, Beerli C, Hofmann A, Hermes E, Muellershausen F, Schubart A, Gardin A. Siponimod (BAF312) penetrates, distributes, and acts in the central nervous system: Preclinical insights. Mult Scler J Exp Transl Clin. 2021 Nov 3;7(4):20552173211049168. doi: 10.1177/20552173211049168. eCollection 2021 Oct. PMID 34777855
- [Background] Berry JD, Paganoni S, Atassi N, Macklin EA, Goyal N, Rivner M, Simpson E, Appel S, Grasso DL, Mejia NI, Mateen F, Gill A, Vieira F, Tassinari V, Perrin S. Phase IIa trial of fingolimod for amyotrophic lateral sclerosis demonstrates acceptable acute safety and tolerability. Muscle Nerve. 2017 Dec;56(6):1077-1084. doi: 10.1002/mus.25733. Epub 2017 Aug 29. PMID 28662296
- [Background] Aytan N, Choi JK, Carreras I, Brinkmann V, Kowall NW, Jenkins BG, Dedeoglu A. Fingolimod modulates multiple neuroinflammatory markers in a mouse model of Alzheimer's disease. Sci Rep. 2016 Apr 27;6:24939. doi: 10.1038/srep24939. PMID 27117087
- See also: Additional citation — https://pubmed.ncbi.nlm.nih.gov/35289055/
- See also: Additional citation — https://www.press.jhu.edu/books/title/12125/fundamental-statistical-methods-analysis-alzheimers-and-other-neurodegenerative